CLINICAL TRIAL: NCT00950209
Title: Acute Effect of Intensive Insulin Infusion on Intestinal Triglyceride-rich-lipoprotein-apoB48 Metabolism in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2007/17; 2007-002791-33
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetic patients in the fed state
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- euglycaemic hyperinsulinic clamp (Active Comparator): In the first step of the protocol, all the patients will have a kinetic study of the TRL-apoB48 in conditions of a saline infusion to measure the "basal" production and clearance rates of the TRL-apoB48. In the second step,the patients of this arm will perform an euglycaemic hyperinsulinic clamp to maintain plasma glucose around 1g/l.
  Interventions: Dietary Supplement: saline infusion; Other: euglycaemic hyperinsulinic clamp
- euglycaemic hyperinsulinic clamp with Endolipide and heparin (Active Comparator): In the first step of the protocol, all the patients will have a kinetic study of the TRL-apoB48 in conditions of a saline infusion to measure the "basal" production and clearance rates of the TRL-apoB48. In the second step,the patients of this arm will perform an euglycaemic hyperinsulinic clamp to maintain plasma glucose around 1g/l but will be also infused with Endolipide 20 % (12,5 ml/h) and heparin (250 U/h) to prevent the suppressive effect of insulin on plasma free fatty acids.
  Interventions: Dietary Supplement: saline infusion; Other: euglycaemic hyperinsulinic clamp; Dietary Supplement: infusion of Endolipide and heparin
- hyperglycaemic hyperinsulinic clamp (Active Comparator): In the first step of the protocol, all the patients will have a kinetic study of the TRL-apoB48 in conditions of a saline infusion to measure the "basal" production and clearance rates of the TRL-apoB48. In the second step,the patients of this arm will perform a hyperglycaemic hyperinsulinic clamp to maintain plasma glucose around 2 g/l to prevent the decreasing effect of insulin on plasma glucose.
  Interventions: Dietary Supplement: saline infusion; Other: hyperglycaemic hyperinsulinic clamp

INTERVENTIONS:
Dietary Supplement: saline infusion — In the first step of the protocol, all the patients will have a kinetic study of the TRL-apoB48 in conditions of a saline infusion to measure the "basal" production and clearance rates of the TRL-apoB48
Other: euglycaemic hyperinsulinic clamp — an euglycaemic hyperinsulinic clamp to maintain plasma glucose around 1g/l
  Arms: euglycaemic hyperinsulinic clamp; euglycaemic hyperinsulinic clamp with Endolipide and heparin
Dietary Supplement: infusion of Endolipide and heparin — an infusion with Endolipide 20 % (12,5 ml/h) and heparin (250 U/h) to prevent the suppressive effect of insulin on plasma free fatty acids
  Arms: euglycaemic hyperinsulinic clamp with Endolipide and heparin
Other: hyperglycaemic hyperinsulinic clamp — a hyperglycaemic hyperinsulinic clamp to maintain plasma glucose around 2 g/l to prevent the decreasing effect of insulin on plasma glucose.
  Arms: hyperglycaemic hyperinsulinic clamp

SUMMARY:
Atherosclerotic cardiovascular disease (ASCD) is the first cause of morbidity and mortality at type 2 diabetes. The typical dyslipidemia that is associated with insulin resistance, which includes a postprandial elevation of triglyceride-rich lipoproteins (TRLs) with excess of intestinal triglyceride-rich-lipoprotein-apoB48 (TRL-apoB48), is felt to play an important role in the accelerated ASCD.

The investigators' objectives in this study are to determine whether an acute elevation of plasma insulin, secondarily to plasma insulin infusion, modulates the production and the clearance rates of intestinal TRL-apoB48 in type 2 diabetic patients in the fed state and to determine if this is a direct effect of insulin or an indirect effect due to the decrease of plasma FFA or the decrease of plasma glucose.

DETAILED DESCRIPTION:
Background: Atherosclerotic cardiovascular disease (ASCD) is the first cause of morbidity and mortality at type 2 diabetes. The typical dyslipidemia that is associated with insulin resistance, which includes a postprandial elevation of triglyceride-rich lipoproteins (TRLs) with excess of intestinal triglyceride-rich-lipoprotein-apoB48 (TRL-apoB48), is felt to play an important role in the accelerated ASCD. Recently, intestinal TRL-apoB48 overproduction appeared as a newly recognized component of insulin resistance. Despite ample evidence supporting the delayed clearance of intestinal TRL-apoB48, there is only a limited amount of information in the literature regarding the factors modulating the production of intestinal TRL-apoB48 in the setting of insulin resistance and type 2 diabetes mellitus. Several arguments suggest that the intestine is not a "passive" organ with respect to lipoprotein production, but an organ metabolically active, receiving information from intestinal lumen and blood and able to modulate its syntheses and its lipid secretions according to the substrata, to the insulin or to other substances. There are functional relationships between the intestine and the liver. For example, it has been recently shown that acute elevation of plasma free fatty acids (FFA) in humans stimulates intestinal TRL-apoB48 and hepatic TRL-apoB100 production.

Aims: Our objectives in this study are to determine whether an acute elevation of plasma insulin, secondarily to plasma insulin infusion, modulates the production and the clearance rates of intestinal TRL-apoB48 in type 2 diabetic patients in the fed state and to determine if this is a direct effect of insuline or an indirect effect due to the decrease of plasma FFA or the decrease of plasma glucose.

Patients and methods: This study will be performed in 30 men with type 2 diabetes in a 2-step protocol. We use a stable isotope method (D3-L-leucine) to study the kinetic of the intestinal TRL-apoB48 and hepatic TRL-apoB100 (production and clearance rates).

In the first step of the protocol, all the patients will have a kinetic study of the TRL-apoB48 in conditions of a saline infusion to measure the "basal" production and clearance rates of the TRL-apoB48. In the second step, type 2 diabetic patients will be divided in 3 different paired groups: one performing an euglycaemic hyperinsulinic clamp to maintain plasma glucose around 1g/l ; one performing an euglycaemic hyperinsulinic clamp to maintain plasma glucose around 1g/l, but being infused with Endolipide 20 % (12,5 ml/h) and heparin (250 U/h) to prevent the suppressive effect of insulin on plasma FFA ; one performing a hyperglycaemic hyperinsulinic clamp to maintain plasma glucose around 2 g/l to prevent the decreasing effect of insulin on plasma glucose.

The research ethics board of the Université de la Méditerranée (Comité de protection des personnes-Sud méditerranée I) and the Afssaps (Agence française de sécurité sanitaire des produits de santé) approved the study and all subjects gave written informed consent prior to their participation.

General objective: Given the potential atherogenicity of the intestinal TRL-apoB48 particles, understanding the factors and the biochemical mechanisms of their accumulation in the plasma in the insulin resistant states may lead to specific therapeutic modalities that reduce their plasma concentration and protect against the highly prevalent atherosclerosis that is associated with insulin resistance and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic patients according to the criteria of the American Diabetes Association
* body mass index between 25 and 40 kg/m2
* Subject the therapeutic care of which bases only on the oral anti-diabetics excepted of glitazones and inhibitors of alpha-glucosidases
* Subject without cardiovascular event in the previous 6 months or perturbing disease the lipid balance assessment (dysthyroidism, pituitary disease, adrenal disease)
* No anemia, no coagulation disturb, creatinine clearance > 60 ml/min, fasting triglycerides < 4g/l

Exclusion Criteria:

* Hypersensitivity to egg
* Subject with severe disease associated with diabete

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To determine whether an acute elevation of plasma insulin, secondarily to plasma insulin infusion, modulates the production and the clearance rates of intestinal TRL-apoB48 in type 2 diabetic patients in the fed state | 3 years

SECONDARY OUTCOMES:
To determine if this is a direct effect of insulin or an indirect effect due to the decrease of plasma FFA or the decrease of plasma glucose. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rene Valero, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique-Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Nogueira JP, Maraninchi M, Beliard S, Padilla N, Duvillard L, Mancini J, Nicolay A, Xiao C, Vialettes B, Lewis GF, Valero R. Absence of acute inhibitory effect of insulin on chylomicron production in type 2 diabetes. Arterioscler Thromb Vasc Biol. 2012 Apr;32(4):1039-44. doi: 10.1161/ATVBAHA.111.242073. Epub 2012 Feb 2. PMID 22308041